CLINICAL TRIAL: NCT01992562
Title: A Phase 4, Randomized, Double-blind, Placebo-controlled, Cross-over Clinical Trial of a Single Shot of Intrathecal Ziconotide for the Treatment of Chronic, Medically Refractory Pain From Painful Peripheral Neuropathy or Myelopathy
Brief Title: Single Shot Intrathecal Ziconotide for Painful Neuropathy or Myelopathy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Logistical issues with study process and recruitment
Sponsor: Aaron Boster (Other)
Responsible Party: Sponsor-Investigator, Aaron Boster, Clinical Neuroimmunologist, OhioHealth
Organization: OhioHealth (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PRIALT01
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Painful Myelopathy; Painful Neuropathy
MeSH Terms: conditions — Neuropathy, Painful | interventions — ziconotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): 5 mcg ziconotide in 1ml of normal saline bolus intrathecal injection
  Interventions: Drug: Ziconotide
- Placebo (Placebo Comparator): 1ml of normal saline bolus intrathecal injection
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Ziconotide
  Other Names: Prialt
  Arms: Treatment
Drug: placebo
  Arms: Placebo

SUMMARY:
This is a phase 4 study being conducted at the Ohio State University Department of Neurology Multiple Sclerosis Research Program. The purpose of the study is to administer a single shot of intrathecal (injection into the space surrounding the spinal cord via a lumbar puncture or spinal tap) ziconotide as a test dose to patients who have chronic painful myelopathy (pain from spinal cord damage) or painful peripheral neuropathy (pain from nerve damage) that has not responded to other pain medicines.

DETAILED DESCRIPTION:
Study Hypothesis: We intend to determine if a single shot trial (SST) of intrathecal (IT) ziconotide will temporarily reduce pain in these patients. In the proposed study, patients will receive two injections, one of which is the ziconotide and one which is a placebo. They will be blinded and not know which order they receive the treatment versus placebo. The results of this clinical trial will provide a focused examination of ziconotide efficacy and safety in patients with painful neuropathies or myelopathies that have not been effectively treated with other pain medications. Moreover, the use of a single shot trial (SST) IT injection in the outpatient setting will provide evidence for application of this technique in outpatient neurological clinical practice, thereby improving access to this specific patient population. Ziconotide is currently FDA approved for this indication and route of administration. Therefore, a study design that improves the feasibility of ziconotide trialing specifically in the neurology clinic (that is, single shot administration) is being used in order to ensure its broader use by neurologists who routinely care for neuropathy and myelopathy patients. Information from this study will also inform future studies of predictors for long term efficacy after pump placement.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women 18 years or older.
2. Neuropathic pain due to peripheral neuropathy or myelopathy
3. Duration of condition greater than 6 months
4. Inadequate control with trials of three or more analgesic agents considered standard care for treatment of neuropathic pain; treatment failure can be either due to lack of efficacy or to intolerable side effects.
5. Documented normal CK and GFR within 6 months preceding screening.
6. Baseline BPI pain severity subscale score of >5/10

Exclusion Criteria:

1. Renal insufficiency
2. History of Myopathy or persistently elevated CK levels
3. History of prior suicide attempt or ideation
4. History of Psychosis
5. Pregnancy or breastfeeding
6. Inability or unwillingness to use contraception
7. Inability to provide consent
8. Inability to tolerate lumbar punctures
9. Receiving systemic anticoagulation therapy (eg. Coumadin)
10. Inability/unwilling to self-catheterize if indicated
11. Change (start, stop, adjust) in home medications 30 days prior to screening visit.
12. Baseline CES-D score > 30
13. Subject has previously failed ziconotide treatment
14. Other factors that in the opinion of the PI would exclude the subject from participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale of Pain Intensity (VASPI) | within 8 hours post injection
  The primary outcome measure of this study is to determine the efficacy of single shot IT ziconotide in treatment of refractory neuropathic pain as a result of painful peripheral neuropathy or myelopathy and to determine the maximal decrease from baseline in VASPI (Visual Analog Scale of Pain Intensity). A responder analysis will also be performed for the VASPI.

SECONDARY OUTCOMES:
Numerical Rating Scale of Pain (NRS) | within 8 hours of Injection
  Used to measure pain intensity on a 0-10 scale.
Brief Pain Inventory (BPI) Scale | within a week of Injection
  Used to assess the severity of pain and the impact of pain on daily functions.
Pittsburgh Sleep Quality Index (PSQI) | within a week of injection
  Used to measure the quality and patterns of sleep in adults.
Patient Global Impression of Change (PGIC) | within 8 hours of injection
  Used to assess the patient's belief about the efficacy of their treatment.

OTHER OUTCOMES:
Timed 25 Foot Walk Test (T25-FW) | within 8 hours of injection
  A quantitative mobility and leg function performance test based on a timed 25-foot walk.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron L Boster, MD, Principal Investigator — OhioHealth
Locations (1):
- The Ohio State University Department of Neurology, Columbus, Ohio, United States